CLINICAL TRIAL: NCT07395570
Title: Efficacy of Computer Aided Detection (CADe) System in Detecting Gastric Neoplasia - a Prospective Tandem Study
Brief Title: Efficacy of CADe System in Detecting Gastric Neoplasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2025.465
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gastric Neoplasia
Keywords: CADe; OIP-Ge1; GC-AI; gastric neoplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CADe System Group (Experimental): During the procedure, the stomach would be examined with the assistance of CADe system by endoscopist.
  Interventions: Device: CADe System

INTERVENTIONS:
Device: CADe System — The endoscopy would be performed using standardized video processing system (EVIS-X1 CV-1500, Olympus Medical Corporations, Tokyo, Japan) and gastroscope (GIF-EZ1500, GIF-XZ1200). A soft black hood (MAJ-1989) would be attached to the distal end of the endoscope. The video processing system would be connected to the OIP-Ge1 (Olympus Medical Corporations, Tokyo, Japan), the novel CADe system, allowing simultaneous artificial intelligence assisted lesion detection, when turned on using conventional white light imaging (WLI).

SUMMARY:
Gastric cancer remains the 5th most common cancers worldwide. It also ranked 5th in the cancer related mortality, causing more than 650'000 deaths per year. Survival of gastric cancer is directly related to the stage of the presentation, with early stage cancers having a significantly better survival. Patients with stage I gastric cancer generally have a 5-year survival of more than 90%. In particular, T1a cancer confined to the mucosa are amenable for endoscopic resection, and patients who underwent such treatment have an excellent survival of 97.2% at 5 years. These patients are not only able to survive longer but also with good quality of life through organ preservation.

However, diagnosis of gastric cancer at an early stage has always been difficult. A meta-analysis of 22 studies from both East and Western population showed a gastric cancer miss rate of 9.4%. Early gastric cancer usually presents with subtle mucosal changes that are hard to detect endoscopically, especially for endoscopists with limited experience in early cancer diagnosis. Background chronic inflammation and high frequency of non-neoplastic lesions often pose significant diagnostic challenges for endoscopists to detect real neoplastic changes. In high incidence countries such as Japan and Korea, the combination of national screening programme as well as good endoscopy training program facilitated high proportion of early gastric cancer detection. Previous studies have showed that significant survival outcome difference between countries with high versus low early cancer detection rate.

Artificial intelligence has emerged as one of the promising technologies that helps enhance endoscopic performance. Numerous high quality randomized studies have demonstrated that computer assisted detection (CADe) system significantly improved colonic adenoma detection rate during screening colonoscopy. Development of gastric cancer CADe system has been much slower than colonic polyp detection. Despite the publication of numerous retrospective studies utilizing endoscopic images in differentiating benign versus malignant gastric lesions, there were only very few completed systems available for clinical real time application. A single centre randomized controlled trial from China demonstrated an improvement in the gastric neoplasm miss rate from 27.3% to 6.1 % when utilizing a novel CADe system.

A novel CADe prototype system (OIP-Ge1, Olympus Medical Corporations, Tokyo, Japan) has recently been developed. The system was developed through collaboration of multiple experts in diagnosing early gastric cancer, collecting more than 100'000 endoscopic images from dozens of high volume centres in Japan. There is currently no prospective clinical data on the actual performance of the prototype CADe system, especially when applied in regions with low proportion of early gastric cancer detection.

The purpose of this study is to investigate the clinical utility of the new CADe system in detection of gastric neoplasia among high risk patients.

If the current study confirms the significant difference in miss rate of gastric neoplasia with the CADe system, a multicentred international randomized controlled trial is planned to compare the efficacy of gastric neoplasia detection with or without the system.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* Deemed at high risk of gastric cancer, defined as below:

  1. Family history of stomach cancer (1st degree relative) for screening, or
  2. Known gastric atrophy/ intestinal metaplasia requiring surveillance, or
  3. Suspicious lesion for repeat diagnostic OGD, or
  4. History of gastric dysplasia / early gastric cancer with endoscopic resection for surveillance
  5. Newly diagnosed early gastric cancer, workup for synchronous cancers

Exclusion Criteria:

* History of gastrectomy (For any reason, including benign and malignant disease)
* Patient who refused to participate
* Patients deemed not fit for consent, including minor patients
* Pregnancy
* Other cases deemed by the examining physician as unsuitable for safe treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with missed gastric neoplasia during first endoscopy without CADe system | 1 day
  Number of patients in whom at least one histologically confirmed gastric neoplasia (Vienna III-V) is not identified during the first endoscopy without CADe, but is identified during the second endoscopy with CADe, divided by the total number of patients undergoing both examinations (unit: %) Miss rate (%) = [Number of patients with ≥1 neoplasia detected only on 2nd endoscopy with CADe] ÷ [Total number of patients undergoing both 1st and 2nd endoscopies] × 100.

SECONDARY OUTCOMES:
Gastric neoplasia detection rate during second endoscopy with CADe System | 1 day
  Suspicious lesion(s) detected would appear as a green box on the main video monitor. Consistent appearance of the green box for more than 2 seconds on the same target area would be considered as a positively detected lesion by the CADe system. Gastric neoplasia detection rate is defined as the gastric neoplasia detection rate during the 2nd endoscopy examination with the assistance of CADe system. (unit: %) Detection rate (%) = [Number of patients with ≥1 neoplasia detected on 2nd endoscopy with CADe] ÷ [Total number of patients undergoing 2nd endoscopy with CADe] × 100.
Time to detect each gastric neoplasia with CADe System | 1 day
  Time in seconds from green box to appear to the stable dentification of a histologically confirmed neoplastic lesion (Vienna III-V), recorded automatically by the CADe system or by time-stamped video review. (unit: second)
Detection rate of non-neoplastic gastric lesions with CADe System | 1 day
  Number of patients in whom at least one endoscopically identified non-neoplastic lesion is detected during the CADe-assisted examination divided by total number of patients undergoing CADe-assisted examination (unit: %).
  Detection rate (%) = [Number of patients with ≥1 non-neoplastic gastric lesion detected] ÷ [Total number of patients examined] × 100.
Miss rate of gastric neoplasia detection with CADe System | 1 day
  Number of patients in whom at least one histologically confirmed gastric neoplasia is visible on the recorded video of the second endoscopy (on retrospective expert review) but is not detected by CADe (no stable box ≥2 seconds), divided by the total number of patients with gastric neoplasia on that second examination (unit: %).
  Miss rate (%) = [Number of patients with ≥1 neoplastic lesion visible on video but not detected by CADe] ÷ [Total number of patients with gastric neoplasia during 2nd endoscopy] × 100.
Total procedure time for screening endoscopy | 1 day
  Time in minutes from scope insertion to scope withdrawal, including the first examination without CADe and the second examination with CADe, measured using the endoscopy unit's time stamps. (unit: minute)
Mean number of lesions detected per endoscopy (neoplastic and non-neoplastic) | 1 day
  Total count of lesions (neoplastic and non-neoplastic) detected during each examination (first without CADe, second with CADe), divided by the number of procedures, reported as mean ± SD per procedure.
  Mean lesions per procedure = [Total number of lesions detected in all procedures] ÷ [Total number of procedures].
Video recording | 1 day
  Digital high-definition video capture system integrated with the endoscopy tower, summarized as percentage of procedures with complete, analyzable recordings. (unit: yes/no, %) Proportion with complete recording (%) = [Number of procedures with complete video adequate for review] ÷ [Total number of procedures] × 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty of Medicine, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Hasuike N, Ono H, Boku N, Mizusawa J, Takizawa K, Fukuda H, Oda I, Doyama H, Kaneko K, Hori S, Iishi H, Kurokawa Y, Muto M; Gastrointestinal Endoscopy Group of Japan Clinical Oncology Group (JCOG-GIESG). A non-randomized confirmatory trial of an expanded indication for endoscopic submucosal dissection for intestinal-type gastric cancer (cT1a): the Japan Clinical Oncology Group study (JCOG0607). Gastric Cancer. 2018 Jan;21(1):114-123. doi: 10.1007/s10120-017-0704-y. Epub 2017 Feb 21. PMID 28224238
- [Background] Pimenta-Melo AR, Monteiro-Soares M, Libanio D, Dinis-Ribeiro M. Missing rate for gastric cancer during upper gastrointestinal endoscopy: a systematic review and meta-analysis. Eur J Gastroenterol Hepatol. 2016 Sep;28(9):1041-9. doi: 10.1097/MEG.0000000000000657. PMID 27148773
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Huang RJ, Koh H, Hwang JH; Summit Leaders. A Summary of the 2020 Gastric Cancer Summit at Stanford University. Gastroenterology. 2020 Oct;159(4):1221-1226. doi: 10.1053/j.gastro.2020.05.100. Epub 2020 Jul 21. PMID 32707045
- [Background] Desai M, Ausk K, Brannan D, Chhabra R, Chan W, Chiorean M, Gross SA, Girotra M, Haber G, Hogan RB, Jacob B, Jonnalagadda S, Iles-Shih L, Kumar N, Law J, Lee L, Lin O, Mizrahi M, Pacheco P, Parasa S, Phan J, Reeves V, Sethi A, Snell D, Underwood J, Venu N, Visrodia K, Wong A, Winn J, Wright CH, Sharma P. Use of a Novel Artificial Intelligence System Leads to the Detection of Significantly Higher Number of Adenomas During Screening and Surveillance Colonoscopy: Results From a Large, Prospective, US Multicenter, Randomized Clinical Trial. Am J Gastroenterol. 2024 Jul 1;119(7):1383-1391. doi: 10.14309/ajg.0000000000002664. Epub 2024 Jan 18. PMID 38235741
- [Background] Gong D, Wu L, Zhang J, Mu G, Shen L, Liu J, Wang Z, Zhou W, An P, Huang X, Jiang X, Li Y, Wan X, Hu S, Chen Y, Hu X, Xu Y, Zhu X, Li S, Yao L, He X, Chen D, Huang L, Wei X, Wang X, Yu H. Detection of colorectal adenomas with a real-time computer-aided system (ENDOANGEL): a randomised controlled study. Lancet Gastroenterol Hepatol. 2020 Apr;5(4):352-361. doi: 10.1016/S2468-1253(19)30413-3. Epub 2020 Jan 22. PMID 31981518
- [Background] Lau LHS, Ho JCL, Lai JCT, Ho AHY, Wu CWK, Lo VWH, Lai CMS, Scheppach MW, Sia F, Ho KHK, Xiao X, Yip TCF, Lam TYT, Kwok HYH, Chan HCH, Lui RN, Chan TT, Wong MTL, Ho MF, Ko RCW, Hon SF, Chu S, Futaba K, Ng SSM, Yip HC, Tang RSY, Wong VWS, Chan FKL, Chiu PWY; ENDOAID-TRAIN study group. Effect of Real-Time Computer-Aided Polyp Detection System (ENDO-AID) on Adenoma Detection in Endoscopists-in-Training: A Randomized Trial. Clin Gastroenterol Hepatol. 2024 Mar;22(3):630-641.e4. doi: 10.1016/j.cgh.2023.10.019. Epub 2023 Nov 2. PMID 37918685
- [Background] Seager A, Sharp L, Neilson LJ, Brand A, Hampton JS, Lee TJW, Evans R, Vale L, Whelpton J, Bestwick N, Rees CJ; COLO-DETECT trial team. Polyp detection with colonoscopy assisted by the GI Genius artificial intelligence endoscopy module compared with standard colonoscopy in routine colonoscopy practice (COLO-DETECT): a multicentre, open-label, parallel-arm, pragmatic randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Oct;9(10):911-923. doi: 10.1016/S2468-1253(24)00161-4. Epub 2024 Aug 14. PMID 39153491
- [Background] Ochiai K, Ozawa T, Shibata J, Ishihara S, Tada T. Current Status of Artificial Intelligence-Based Computer-Assisted Diagnosis Systems for Gastric Cancer in Endoscopy. Diagnostics (Basel). 2022 Dec 13;12(12):3153. doi: 10.3390/diagnostics12123153. PMID 36553160
- [Background] Wu L, Shang R, Sharma P, Zhou W, Liu J, Yao L, Dong Z, Yuan J, Zeng Z, Yu Y, He C, Xiong Q, Li Y, Deng Y, Cao Z, Huang C, Zhou R, Li H, Hu G, Chen Y, Wang Y, He X, Zhu Y, Yu H. Effect of a deep learning-based system on the miss rate of gastric neoplasms during upper gastrointestinal endoscopy: a single-centre, tandem, randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Sep;6(9):700-708. doi: 10.1016/S2468-1253(21)00216-8. Epub 2021 Jul 21. PMID 34297944
- [Background] Yao K. The endoscopic diagnosis of early gastric cancer. Ann Gastroenterol. 2013;26(1):11-22. PMID 24714327
- [Background] Muto M, Yao K, Kaise M, Kato M, Uedo N, Yagi K, Tajiri H. Magnifying endoscopy simple diagnostic algorithm for early gastric cancer (MESDA-G). Dig Endosc. 2016 May;28(4):379-393. doi: 10.1111/den.12638. Epub 2016 Apr 22. PMID 26896760